CLINICAL TRIAL: NCT05726188
Title: Predictors of Disease Recurrence After Curative Surgery for Stage I Colon Cancer - CORE1 (COlon Cancer REcurrence in Stage 1)
Brief Title: Predictors of Disease Recurrence After Curative Surgery for Stage I Colon Cancer
Acronym: CORE1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: CORE1
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Colon Cancer Stage I; Colon Cancer
Keywords: prognosis; recurrence
MeSH Terms: conditions — Colonic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage I colon cancer: Patients aged 18 years or above with pT1 or pT2 N0 colon cancer (up to the recto-sigmoid junction) who underwent curative resection between January 2010 and December 2019
  Interventions: Procedure: Colonic resection

INTERVENTIONS:
Procedure: Colonic resection — Elective or urgent colonic resection; minimally-invasive or open surgery; completion surgery for endoscopically resected pT1 colon cancer with high risk features

SUMMARY:
Patients with stage I (pT1-2 N0 M0) colon cancer (CC) accounts for 15-20% of colonic neoplasia. Stage I CC is mostly cured with surgical resection, consequently, adjuvant chemotherapy is never considered for this subset of patients. Moreover, some international guidelines, including NCCN guidelines, recommend less intensive follow-up 1. However, around 5% of patients with stage I CC will develop a recurrence within 5 years from surgery. Despite the very good prognosis usually attributed to this stage (5-years relapse-free survival: 95%), some clinical and pathological factors beyond the standard AJCC staging may be associated with worse clinical features and may aid in prognostic stratification. Although some authors investigated the role of pathological and clinical factors in patients with stage II and III disease, only few data are available for patients with stage I CC1.

The present multicentric retrospective study aims to:

1. Assess the actual incidence of recurrence in a large cohort of patients with stage I CC undergone curative resection.
2. Investigate the clinical and pathological characteristics of patients who developed a recurrence, with the aim of identifying those associated with a significantly increased risk.
3. Analyze the pattern of recurrence.
4. Analyze survival after recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Colon cancer up to recto-sigmoid junction
* Histological diagnosis of adenocarcinoma
* pT1 or pT2 according to AJCC staging system
* Urgent and elective surgery
* Curative resection
* Minimally invasive or open surgery
* Completion surgery included (Surgery for endoscopically resected pT1)

Exclusion Criteria:

* Rectal cancer
* Adenoma with low- or high-grade dysplasia
* Histology other than adenocarcinoma (i.e., lymphoma, neuroendocrine tumor, squamous carcinoma, etc)
* Neo-adjuvant chemotherapy or radiotherapy
* History of tumors other than CC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I colon cancer who underwent curative surgery at the participating centers between January 2010 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 5 years
  Number of patients who relapsed after curative resection

SECONDARY OUTCOMES:
Overall survival | 5 years
  Percentage of patients alive 5 years after surgery
Cancer-related survival | 5 years
  Percentage of patients who did not die from cancer-related causes

CONTACTS AND LOCATIONS:
Locations (24):
- Unit of Digestive and HPB Surgery, Henri Mordor University Hospital, Paris, France
- Italy (23):
  - Chirurgia dell'Apparato Digerente, IRCSS Giovanni Paolo II, Bari
  - Chirurgia Generale e Trapianto di Fegato, Azienda Ospedaliera Consorziale Policlinico di Bari, Bari
  - UO Chirurgia Generale 3, Spedali Civili 1, Brescia
  - Chirurgia Coloproctologica, AOU Cagliari, Cagliari
  - Chirurgia Generale, Ospedale di Cles, Cles
  - Chirurgia 1, Ospedale di Cona, AOUI Ferrara, Cona
  - Chirurgia Generale Colorettale, Ospedale degli Infermi, Faenza
  - UOS Chirurgia Colo-rettale, Ospedale San Gerardo, Monza
  - Chirurgia Endoscopica, AOUI Federico II, Napoli
  - UOC Oncologia Chirurgia Colorettale, Istituto Nazionale Tumori - IRCCS Fondazione Pascale, Napoli
  - Chirurgia Generale, AOU San Luigi Gonzaga, Orbassano
  - Chirurgia Generale 3, AOUI Padova, Padua
  - ASL TO 3 Presidio Pinerolo, Chirurgia, Pinerolo
  - Chirurgia Generale 2, Policlinico Gemelli, Roma
  - Policlinico TOR Vergata, Roma, Chirurgia Mininvasiva e dell'Apparato Digerente, Roma
  - UOC Chirurgia Generale 1, Policlinico Gemelli, Roma
  - Chirurgia Generale, Ospedale Santa Maria della Misericordia, Rovigo
  - Chirurgia Colorettale, IRCCS Humanitas, Rozzano
  - Chirurgia d'Urgenza e PS 3, AOU Città della Salute e della Scienza, Torino
  - Chirurgia Generale e Mininvasiva, Ospedale San Camillo, Trento
  - SC Clinica Chirurgia, Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
  - Unità di Chirurgia Colorettale, Clinica Santa Rita, Vercelli
  - Chirurgia Generale ed Epatobiliare, AOUI Verona, Verona

IPD SHARING:
Plan to Share IPD: No